CLINICAL TRIAL: NCT02832882
Title: Radiofrequency Ablation for Small Hepatocellular Carcinoma Using Octopus Electrode and No-touch Technique: Preliminary Study
Brief Title: RFA for Small HCC With No-touch Technique Using Octopus Electrode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUH-2016-2244
Record Dates: First submitted 2016-06-03; First posted 2016-07-14 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; RFA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No-touch RFA arm (Experimental): No-touch RFA arm indicates RFA procedure using Octopus electrode and no touch technique.
  Interventions: Procedure: No-touch RFA
- Conventional tumor puncture RFA arm (Active Comparator): Conventional tumor puncture RFA arm indicates RFA procedure using Octopus electrode and conventional tumor puncture technique.
  Interventions: Procedure: Conventional tumor puncture RFA

INTERVENTIONS:
Procedure: No-touch RFA — No-touch RFA indicates RFA without tumor puncture. In this study, no-touch RFA is performed using Octopus electrodes.
  Arms: No-touch RFA arm
Procedure: Conventional tumor puncture RFA — Conventional tumor puncture RFA indicates routine procedure of RFA in our institution. In this study, RFA procedure is performed using Octopus electrodes.
  Arms: Conventional tumor puncture RFA arm

SUMMARY:
In this study, the investigators are going to prospectively compare the clinical outcomes (technical success rate, 12 month local tumor progression rate, complication rate, tumor seeding rate) of Radiofrequency ablation (RFA) with octopus electrode and no-touch technique for Hepatocellular carcinoma (HCC) to those of RFA with conventional tumor puncture method with the same device.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh class A
* patient with 1cm-2.5cm sized HCC
* 1 or 2 HCCs
* being referred for curative purpose of RFA
* sign informed consent

Exclusion Criteria:

* maximum tumor diameter greater than 2.5cm
* Child-Pugh class B or C
* more than 3 HCC lesions
* invisible tumor even after US/CT or US/MR fusion
* presence of vascular tumor thrombosis or extrahepatic metastasis
* severe coagulopathy (PLT < 50K, PT < 50% of normal range)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
12 month local tumor progression (LTP) rate | 12 month after RFA

SECONDARY OUTCOMES:
tumor seeding rate | 12 months after RFA
  incidence of tract seeding after RFA.
Complication rate related with RFA | 1 month
  RFA-related complication rate such as death, abscess, bleeding..etc.
Technical success rate | 1 months
  presence or absence of residual lesion on follow-up imaging

OTHER OUTCOMES:
Ablation time | 3 days after RFA
  ablation time for tumor ablation
Intrahepatic distant mets | 12 months after RFA
  incidence of intrahepatic distant metastasis after RFA
Extrahepatic distant mets | 12 months after RFA
  incidence of extrahepatic distant metastasis after RFA
Technical efficacy 1 | 2 days after RFA
  Assessment of ablative margin using score 1-4 (1: residual tumor; 4: equal to or larger than 5mm) in side-by-side comparison of pre-RFA CT/MR and post-RFA CT using visual assessment
Technical efficacy 2 | 2 days after RFA
  Assessment of ablative margin using score 1-4 (1: residual tumor; 4: equal to or larger than 5mm) in side-by-side comparison of pre-RFA CT/MR and post-RFA CT using registration software

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No